CLINICAL TRIAL: NCT06712121
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy of VEnetoclax and DEciTabine in Relapsed/Refractory Adult T-acute Lymphoblastic lEukemia/Lymphoma
Brief Title: Venetoclax and Decitabine in R/R T-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Society of Hematology (Network)
Responsible Party: Principal Investigator, Dong-Yeop Shin, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEDETTE
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma
Keywords: T lymphoblastic leukemia/lymphoma; venetoclax; decitabine
MeSH Terms: conditions — Lymphoma | interventions — Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- decitabine and venetoclax arm (Experimental): arm treated with venetoclax plus decitabine
  Interventions: Drug: decitabine plus venetoclax

INTERVENTIONS:
Drug: decitabine plus venetoclax — decitabine 20mg/m2 for 7 days venetoclax 400mg daily for 21 days

SUMMARY:
The goal of this phase 2 clinical trial is to test the efficacy of decitabine and venetoclax combination chemotherapy in relapsed or refractory adult T-cell acute lymphoblastic leukemia/lymphoblastic lymphoma.

This study use a modified regimen of decitabine and venetoclax.

DETAILED DESCRIPTION:
Our study is conducted in collaboration with Korean adult acute lymphoblastic leukemia working party (KALLWP) and consortium for improving survival of lymphoma (CISL). This study recruits adult patients with R/R T-ALL/LBL and treated with 7-day decitabine plus 3 weeks of venetoclax up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older but less than 80 years
* Eastern Cooperative Oncology Group Performance Score (ECOG PS) ≤ 2
* Confirmed diagnosis of T-cell lymphoblastic leukemia/lymphoma according to the 2016 World Health Organization criteria, with relapse or failure to achieve complete remission despite induction chemotherapy
* Patients with peripheral blood leukocytes <50,000/uL (reducing white blood cell count through hydroxyurea or leukapheresis prior to trial enrollment is allowed)
* At the time of screening, a calculated glomerular filtration rate (GFR) ≥ 30 mL/min according to the Cockcroft-Gault formulas, or creatinine ≤ 1.4, total bilirubin ≤ 3.0 mg/dL, and AST and ALT < x5 upper limit of normal (ULN) (however, if bilirubin elevation is due to Gilbert's syndrome or liver enzyme elevation is due to infiltration of leukemia/lymphoma, enrollment may be allowed even if the above conditions are exceeded)
* Individuals who agree to the following contraceptive measures for a period of 3 months during treatment and for 3 months after completion:

Exclusion Criteria:

* Individuals in complete remission with previous treatment, if relapse or resistance is not confirmed by bone marrow examination or imaging/tissue examination.
* Individuals who previously received venetoclax + decitabine treatment for T-lymphoblastic leukemia/lymphoma (participants who received venetoclax + decitabine treatment for a different type of cancer [e.g., acute myeloid leukemia] and have elapsed more than 1 year since the last treatment are allowed).
* Pregnant or breastfeeding individuals.
* Individuals who received systemic anticancer chemotherapy or participated in a clinical trial treatment within the past 2 weeks.
* Individuals with active leukemia involving the central nervous system.
* Individuals with a cancer type other than T-lymphoblastic leukemia/lymphoma that requires current active treatment (participants with a cancer type that has already been cured or is in a slow-progressing state without treatment, as determined by surgery/radiation/chemotherapy, may participate under the consultation of the clinical trial investigator).
* Individuals with active human immunodeficiency virus (HIV) infection, hepatitis B/hepatitis C infection (participants without evidence of viral particles through PCR testing may be enrolled with the consent of an infectious disease specialist or hepatologist).
* Uncontrolled bleeding.
* Uncontrolled infection (bacterial, fungal, viral).
* Uncontrolled mental illness.
* Individuals who do not understand the informed consent or have difficulty in adequate communication, making them inappropriate for participation in the clinical trial.
* Cases where the investigator judges that patient evaluation may be hindered or participation in the clinical trial is not appropriate.
* Individuals who have a negative attitude towards participating in the clinical trial or who are unwilling to comply with the treatment and specimen collection schedule specified in the study protocol.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The rate of composite Complete remission | 1 year
  CR: complete remission CRh: complete remission with partial hematologic recovery CRi: complete remission with incomplete hematologic recovery MLFS: morphologic leukemia-free state

SECONDARY OUTCOMES:
Composite overall response rate | 1 year
  cORR: CR/CRh/CRi/MLFS+PR
Clinical benefit rate | 1 year
  CR: complete remission CRh: complete remission with partial hematologic recovery CRi: complete remission with incomplete hematologic recovery MLFS: morphologic leukemia-free state PR: partial remission stable disease
Duration of response | 1 year
  by months
Bridging to allogeneic hematopoietic stem cell transplantation (HSCT) | 1 year
  by rate
Progression-free survival (PFS) | 1 year
  by months
Overall survival (OS) | 1 year
  by months

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No